CLINICAL TRIAL: NCT03872258
Title: Effectiveness of an Intensive Intervention to Improve Physical Activity in Postmenopausal and Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRS 1823/B/18
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Physical activity; Postmenopause; Body composition; Health education; Information and Communication Technologies
MeSH Terms: conditions — Motor Activity; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Counseling on physical activity
  Interventions: Behavioral: Control
- Intervention (Experimental): Add an intensive program of combined exercise for 6 months and use during this period a Smartband, in order to encourage and increase physical activity and decrease sedentary lifestyle
  Interventions: Behavioral: Control; Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Control — Counseling on physical activity
Behavioral: Intervention group — Program of combined exercise and a Smartband for 6 months.
  Arms: Intervention

SUMMARY:
This is a randomized clinical trial aimed at postmenopausal women aged 45 to 70 years old selected in urban primary care centers of two centers (Spain). Its objective is to evaluate the effects of an intensive intervention in the increase of physical activity and the decrease of sedentary lifestyle in postmenopausal and sedentary women.

DETAILED DESCRIPTION:
Objective: to evaluate the effects at 6 months of an intensive intervention in the increase of physical activity and the decrease of sedentary lifestyle in postmenopausal and sedentary women.

Design and setting: A randomized clinical trial of two parallel groups. Population: 100 postmenopausal women, 45 to 70 aged will be included, selected by consecutive sampling in two primary care centers.

Measurements and intervention: Physical activity, body composition, BMI and health-related quality of life will be evaluated. The intervention group will receive an intensive program of combined exercise for 6 months and use during this period a Smartband, in order to encourage and increase physical activity and decrease sedentary lifestyle

ELIGIBILITY:
Inclusion Criteria:

* Women in postmenopausal period defined as 12 consecutive months of amenorrhea.

Exclusion Criteria:

* Older than 70 years are excluded, due to difficulties in the use of Information and Communication Technologies.
* History of cardiovascular events (acute myocardial infarction, stroke, etc).
* Diagnosis of clinically demonstrable neurological and/or neuropsychological disease.
* Muscular-skeletal pathology that inhibit mobility.
* Those with any other circumstance that the investigators consider could interfere with the study procedures.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Physical activity | 6 months
  Physical activity, will be measured using an accelerometer
Self-reported physical activity | 6 months
  Measured by the International Physical Activity Questionary - Short Form
Self-reported sedentary | 6 months
  Measured by the Marshall Questionary

SECONDARY OUTCOMES:
Body composition | 6 months
  Measurement by InBody 230.
Body mass index | 6 months
  Measurement by InBody 230

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia-Ortiz, Study Chair — Primary Health Care Research Unit, The A
Locations (1):
- Instituto Biosanitario de Salamanca. Research unit La Alamedilla, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alonso-Dominguez R, Sanchez-Aguadero N, Llamas-Ramos I, Lugones-Sanchez C, Gonzalez-Sanchez S, Gomez-Marcos MA, Garcia-Ortiz L; Ewomen Investigators. Effect of an intensive intervention on the increase of physical activity and the decrease of sedentary lifestyle in inactive postmenopausal. J Adv Nurs. 2021 Apr;77(4):2064-2072. doi: 10.1111/jan.14737. Epub 2021 Jan 22. PMID 33481300